CLINICAL TRIAL: NCT06307639
Title: Seminal Levels of PGK2 and ACRV1 as Predictors of Micro-TESE Results in NOA
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Muhammad Yousef Muhammad Swifee, Assistant lecturer of Andrology ,Sexology and STIs, Assiut University
Other Study IDs: MYMSwifee
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Male Infertility Due to Azoospermia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measurement of PGK2 and ACRV1 levels in the semen of infertile males undergoing testicular sperm extraction (TESE). — Measurement of PGK2 and ACRV1 levels in the semen of infertile males undergoing testicular sperm extraction (TESE).

SUMMARY:
* Measurement of PGK2 and ACRV1 levels in the semen of infertile males undergoing testicular sperm extraction (TESE).
* Correlate seminal levels of PGK2 and ACRV1 with sperm retrieval results and histopathology analysis of testicular biopsy samples.

ELIGIBILITY:
Inclusion Criteria:

* Infertile males with normal volume, functional (non-obstructive) azoospermia.
* Age: 18-45 years

Exclusion Criteria:

* Patients with proven obstructive azoospermia.
* Cryptorchidism.
* Testicular Agenesis and testicular atrophy.
* Patient with exposure to gonadal toxins like chemotherapy, radiotherapy, and alkylating agents.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Infertile males with normal volume, functional (non-obstructive) azoospermia.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Know more about the functional role of PGK2 and ACRV1 in the process of spermatogenesis. | 2 years
Detect if PGK2 and/or AVRV1 level can used as predictor for spermatogenesis in infertile men with non-obstructive azoospermia undergoing Testicular Sperm Extraction. | 2 years

IPD SHARING:
Plan to Share IPD: No